CLINICAL TRIAL: NCT02470182
Title: Screening for Sleep Disordered Breathing With Minimally Obtrusive Sensors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brian R Snider, Ph.D. Candidate, Oregon Health and Science University
Other Study IDs: IRB00010124
Record Dates: First submitted 2015-05-26; First posted 2015-06-12 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea Syndromes; Snoring
Keywords: sleep apnea; snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- At-Home: Overnight sleep at home (30 subjects)
- Sleep Lab: Overnight sleep at the OHSU sleep lab during routine polysomnography (30 subjects)
- Sleep Lab + At-Home: Overnight sleep at the OHSU sleep lab during routine polysomnography, followed by overnight sleep at home (30 subjects)

SUMMARY:
The purpose of this study is to learn more about breathing disorders during sleep. The investigators want to learn how breathing sounds made during sleep relate to breathing disorders during sleep.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility of assessing breathing problems during sleep with minimally obtrusive sensors (a bedside microphone and wireless pulse oximeter worn on the fingertip). The investigators will use the data collected with these sensors to develop algorithms for automatically detecting sleep apnea events. Subjects will be asked to place unobtrusive sensors (bedside microphone and wireless pulse oximeter) in their home sleep environment. The subjects will start the at-home data collection before they fall asleep, and stop the data collection the next morning when they wake. The subjects will then return the sensors to the investigator for analysis.

We are looking for people interested in participating in the at-home portion of our study. We will only collect at-home data for one night of sleep per subject. After this one night, no further data collection or monitoring will occur. Subjects will be compensated for their time.

A standard sleep-breathing questionnaire (the "Berlin Questionnaire") will be administered. This questionnaire is widely used as a screening tool to determine if a person may have disordered breathing during sleep. This questionnaire consists of 10 multiple-choice questions related to snoring, daytime sleepiness, and other related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-89
* No self-reported sleep breathing problems

Exclusion Criteria:

* Prior diagnosis for a sleep breathing problem (such as sleep apnea)
* Self-reported insomnia
* History of stroke
* Nasal or soft palate surgery in the last 12 months
* Use of a breathing assistance device (such as a CPAP machine)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants must be age 21-89 and have no self-reported sleep breathing problems. Participants must not use a breathing assistance device (such as a continuous positive airway pressure, or CPAP, machine) during sleep.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Non-typical breathing sounds or patterns correspond to oxygen desaturation | On the day of the study only (1 day)
  This study aims to see if it is feasible to assess breathing problems during sleep using a high-quality microphone and wireless pulse oximeter. Our primary objective is to determine if non-typical breathing sounds or patterns correspond to oxygen desaturations of 3% or more from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jan van Santen, Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Center for Spoken Language Understanding, Portland, Oregon, United States